CLINICAL TRIAL: NCT01541774
Title: A Prospective, Multicenter Clinical Evaluation of the Safety and Effectiveness of the Phoenix Atherectomy™ System in Atherectomy of the Peripheral Vasculature
Brief Title: Endovascular Atherectomy Safety and Effectiveness Study
Acronym: EASE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AtheroMed, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP0782
Record Dates: First submitted 2010-08-04; First posted 2012-03-01 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Peripheral Vascular Disease
Keywords: Atherectomy; Atherosclerosis; Peripheral artery disease
MeSH Terms: conditions — Peripheral Vascular Diseases; Atherosclerosis; Peripheral Arterial Disease | interventions — Atherectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Phoenix Atherectomy System (Experimental)
  Interventions: Device: Phoenix Atherectomy System

INTERVENTIONS:
Device: Phoenix Atherectomy System — Evaluate the procedural safety and effectiveness of the Phoenix Atherectomy™ System for the treatment of de novo and restenotic atherosclerotic lesions located in native peripheral arteries as assessed through 30 day follow-up. Further evaluations of device performance ensuring no prostenotic response as assessed through six month follow-up.
  Other Names: Atherectomy; Percutaneous Transluminal Atherectomy; Transluminal Atherectomy; Percutaneous Atherectomy

SUMMARY:
The purpose of this study is to evaluate the procedural safety and effectiveness of the Phoenix Atherectomy™ System for the treatment of de novo and restenotic atherosclerotic lesions located in the native peripheral arteries. The Phoenix Atherectomy™ System is intended for use in atherectomy of the peripheral vasculature. The intended peripheral vessels include the Superficial Femoral, Popliteal, and Infrapopliteal arteries. The system is not intended for use in the coronary, carotid, iliac or renal vasculature. The results of this study will be used to support a 510(k) submission to the Food and Drug Administration.

ELIGIBILITY:
Inclusion Criteria:

* Subject willing and able to give informed consent
* Subject willing and able to comply with the study protocol
* Age ≥18 years old
* Objective hemodynamic criteria that subject has a resting ankle-brachial index (ABI) ≤ 0.90, or ≤ 0.75 after exercise, OR patients with non-compressible arteries (ABI>1.1) must have a toe-brachial index (TBI) of ≤ 0.80
* Clinical description of lesion as characterized by a Rutherford Clinical Class 2 to 5
* Subject is a suitable candidate for angiography and endovascular intervention in the opinion of the investigator or per hospital guideline
* Subject has target lesion/lesions defined as stenosis ≥ 70% as determined by operator visual assessment, distal to the profunda femoral artery. No more than two lesions may be treated with the Phoenix device and one of the treated lesions must include a lesion with the worst percent diameter stenosis.
* Total treated lesion length with the Phoenix device ≤ 10 cm
* Popliteal and above, target reference vessel diameter (proximal and distal to target lesion) is ≥ 2.5 mm and ≤ 4.5 mm
* At least one patent tibial vessel runoff at baseline.
* Below popliteal, target reference vessel diameter (proximal and distal to target lesion) is ≥ 2.5 mm and ≤ 3.5 mm

Exclusion Criteria:

* Patient has an active infection in the target limb
* Clinical/angiographic complication (other than non-flow limiting dissections) attributed to a currently marketed device prior to introduction of Phoenix System
* Critical limb ischemia with Rutherford Clinical Class 6
* Target lesion containing severe calcification that is circumferential and noted in two views
* Lesion in the contralateral limb requiring intervention during index procedure or within next 30 days
* In-stent restenosis within the target lesion
* Flow limiting dissection, Type C or greater
* Lesion within a native vessel graft or synthetic graft
* History of an endovascular procedure or open vascular surgery on the index limb within the last 30 days
* Subject has any planned surgical or interventional procedure within 30 days after the study procedure
* Significant acute or chronic kidney disease with a creatinine level >2.5 mg/dl, and/or requiring dialysis
* Unstable coronary artery disease or other uncontrolled comorbidity
* Myocardial infarction or stroke within 2 months of baseline evaluation
* Subject is pregnant or breast-feeding
* Participation in any study of an investigational device, medication, biologic, or other agent within 30 days prior to enrollment that is either a cardiovascular study or could, in the judgment of the investigator, affect the results of this study
* Subject has significant stenosis or occlusion of inflow tract (upstream disease) not successfully treated before this procedure
* Subject in whom antiplatelet, anticoagulant, or thrombolytic therapy is contraindicated
* Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 125,000/microliter, known coagulopathy, or INR > 1.5
* Known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated
* History of heparin-induced thrombocytopenia (HIT)
* Any thrombolytic therapy within two weeks of enrollment
* Psychiatric disorder which in the judgment of the investigator could interfere with provision of informed consent, completion of tests, therapy, or follow-up
* Clinical/angiographic evidence of distal embolization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2010-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety: Freedom from Major Adverse Events | 30 days
Efficacy: Technical Success | Day 1
  The achievement of acute debulking to achieve a post-Phoenix (prior to any adjunctive therapy) residual diameter stenosis of ≤50%.

SECONDARY OUTCOMES:
Assessment of Major Adverse Events | From 1 month to 6 months post procedure
Procedural success | Day 1
  Procedural success rate is defined as the proportion of the target lesions in which the final stenosis is <30% after treatment with atherectomy and any other adjunctive therapy.
Clinical success | 30 days to 6 months
  Clinical success rate is defined as the proportion of subjects that have procedural successes in all target lesions with achievement of at least one Rutherford Clinical Scale at 30 days and 6 months post procedure,
Target vessel Revascularization | Treatment through 6 months
  Incidence of clinically-driven target vessel revascularization or target limb revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Davis, MD, Principal Investigator — St. John Hospital & Medical Center; James McKinsey, MD, Principal Investigator — Columbia University Medical Center/New York Presbyterian
Locations (16):
- United States (14):
  - Spring Hill Medical Center, Mobile, Alabama
  - Arizona Heart Institute, Phoenix, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Vascular Interventional Center, Pensacola, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - WellStar Health System, Austell, Georgia
  - Methodist Research Imstitute /Cobb Hospital, Indianapolis, Indiana
  - Cardiovascular Institute of the South, Houma, Louisiana
  - Cardiovascular Inst The Regional Med Center/Center of Acadia Institute of the South, Lafayette, Louisiana
  - St. John Hospital and Medical Center, Detroit, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Hunterdon Cardiovascular Associated, Flemington, New Jersey
  - Columbia University Medical Center/New York Presbyterian, New York, New York
  - The Carl & Eduth Lindner Center for Research & Education at the Christ Hospital, Kingsport, Tennessee
- Germany (2):
  - Hochrhein-Eggberg-Klinik GmbH, Bad Säckingen, Germany
  - Park-Hospital Leipzig, Leipzig, Germany

REFERENCES:
- [Derived] Davis T, Ramaiah V, Niazi K, Martin Gissler H, Crabtree T. Safety and effectiveness of the Phoenix Atherectomy System in lower extremity arteries: Early and midterm outcomes from the prospective multicenter EASE study. Vascular. 2017 Dec;25(6):563-575. doi: 10.1177/1708538117712383. Epub 2017 Sep 27. PMID 28950783